CLINICAL TRIAL: NCT05374694
Title: Epigenetic Characterization of Angina Pectoris According to the Affected Coronary Compartment: Relationship Between Invasive Physiological Coronary Evaluation and Micro-RNAs
Brief Title: Angina, Physiology, Biology (ANgina, FIsiologia BIOlogia)
Acronym: ANFIBIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Arnau de Vilanova (Other)
Responsible Party: Principal Investigator, Diego Fernández-Rodríguez, Principal Investigator, Hospital Arnau de Vilanova
Other Study IDs: CEIC-2665
Record Dates: First submitted 2022-05-05; First posted 2022-05-16 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Angina Pectoris
Keywords: Coronary physiology; Biology; miRNA; Fractional flow reserve; Index of microcirculatory resistance; Angina pectoris
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Overexpression in angina: miR-1-3p, miR-21-5p, miR-133a-3p, miR-133b-3p, miR-208a-3p, miR-208b-3p, miR-125a-5p, miR-187-3p , miR-499a-5p, miR-502-5p.
  * Underexpression in angina: miR-100-5p, miR-143-3p, miR-145-3p, miR-29b-5p. Open to explore other micro-RNAs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1: Macrovasculature + (FFR ≤ 0.80) / Microvasculature + (IMR ≥25)
  Interventions: Diagnostic Test: Physiological invasive coronary evaluation
- Group 2: Macrovasculature + (FFR ≤ 0.80) / Microvasculature - (IMR <25)
  Interventions: Diagnostic Test: Physiological invasive coronary evaluation
- Group 3: Macrovasculature - (FFR>0.80) / Microvasculature + (IMR ≥25)
  Interventions: Diagnostic Test: Physiological invasive coronary evaluation
- Group 4: Macrovasculature - (FFR>0.80) / Microvasculature - (IMR <25)
  Interventions: Diagnostic Test: Physiological invasive coronary evaluation
- Group 5: Microvascular spasm (<90% diameter contraction, Chest pain, ECG changes) or Macrovascular spasm (>90% diameter contraction, Chest pain, ECG changes)
  *Only patients in groups 3 and 4 will undergo the acetylcholine test.
  Interventions: Diagnostic Test: Physiological invasive coronary evaluation

INTERVENTIONS:
Diagnostic Test: Physiological invasive coronary evaluation — Performance of FFR, IMR and acetylcholine test (Only patients in groups 3 and 4 will undergo the acetylcholine test)

SUMMARY:
Relationship between invasive physiological assessment with FFR and IMR and biological markers as micro-RNA's according to coronary vascular compartiment affected (Group 1: Macrovasculature + / Microvasculature +; Group 2: Macrovasculature + / Microvasculature -; Group 3: Macrovasculature - / Microvasculature +; Group 4: Macrovasculature - / Microvasculature -). Also, biological markers will be related with presence of microvascular spasm or macrovascular spasm (Group 5).

DETAILED DESCRIPTION:
Patients with chest pain suggestive of angina after ruling out other cardiac and non-cardiac causes, referred for invasive coronary angiography, will be evaluated by coronary angiography and invasive coronary physiological assessment by determining FFR and IMR and by performing a vasoreactivity test with acetylcholine.

A relationship will be established between the invasive physiological assessment with FFR and IMR and biological markers such as micro-RNA's according to the affected coronary vascular compartment (Group 1: Macrovasculature + / Microvasculature +; Group 2: Macrovasculature + / Microvasculature -; Group 3 : Macrovasculature - / Microvasculature +; Group 4: Macrovasculature - / Microvasculature -). In addition, the biological markers will be related to the presence of microvascular spasm or macrovascular spasm (Group 5).

Finally, among other biological markers, the following miRNAs will be compared. These miRNA's present consistent data in the literature about their over or underexpression.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients with chest pain suggestive of angina evaluated by a cardiologist referred for diagnostic coronary angiography and possible coronary intervention.
3. Echocardiogram ruling out noncoronary cardiac causes of chest pain.
4. Informed consent.

Exclusion Criteria:

1. Contrast allergy not susceptible to premedication.
2. Severe bronchial asthma or adenosine intolerance.
3. Atrio-ventricular block (≥ 2nd degree) or acetylcholine intolerance.
4. Acute myocardial infarction with ST-segment elevation.
5. Acute myocardial infarction without ST-segment elevation.
6. Cardiogenic shock.
7. Total occlusion of any coronary artery that precludes measurements with pressure-temperature guidewires.
8. Previous coronary artery bypass grafting.
9. Women with the possibility of being pregnant.
10. Renal dysfunction with an estimated glomerular filtration rate <30 mL/min/1.73m2.
11. Inability to understand the nature of the study and / or sign informed consent.
12. Any other medical condition that, in the opinion of the researcher, may lead to safety issues for patients or may alter the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with angor pectoris referred for coronary angiography after excluding other cardiaca and non-cardiac causes of chest pain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
FFR | Intraprocedure
  Fractional flow reserve
IMR | Intraprocedure
  Index of microvascular resistance
Ach | Intraprocedure
  Acetilcholine test

SECONDARY OUTCOMES:
QCA | Intraprocedure
  Quantitative Coronary Angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Arnau de Vilanova, Lleida, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: No specific time frame
Access Criteria: Each center will fill an anonymized and predefined case report form (CRF) developed by the investigators. The selected variables are oriented to the cardiovascular risk factors, comorbidities, clinical findings, ischemia detection tests, medications, analytical parameters, echocardiographic and angiographic findings, and invasive physiological indexes. All data collected during the study, after deidentification, will be shared. Data obtained through this study may be provided to qualified researchers with academic interest in cardiovascular diseases. Approval of the request and execution of all applicable agreements are prerequisites for the sharing of data with the requesting party.